CLINICAL TRIAL: NCT01590446
Title: A Phase 1, Two-Part, Double-Blind, Placebo-Controlled Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of BMN 111 Administered to Healthy Adult Volunteers
Brief Title: A Study to Evaluate Safety and Tolerability of BMN 111 Administered to Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 111-101
Record Dates: First submitted 2012-03-14; First posted 2012-05-03 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Achondroplasia
Keywords: Achondroplasia
MeSH Terms: conditions — Achondroplasia | interventions — vosoritide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Normal Saline
- BMN 111 (Active Comparator)
  Interventions: Drug: BMN 111

INTERVENTIONS:
Drug: BMN 111 — SC injection, Part 1 single dose and Part 2 multiple dose.
  Other Names: Modified C-Natriuretic Peptide, ProCNP38
  Arms: BMN 111
Drug: Normal Saline — SC injection, Part 1 single dose and Part 2 multiple dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure how much of the study drug gets into the blood- stream and how long it takes the body to get rid of it when given as a single dose. Information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to provide written, signed informed consent (legally authorized representative) after the nature of the study has been explained and prior to performance of any research-related procedure.
* Is a male 22 to 45 years of age, inclusive
* Has a body weight between 63 and 100 kg, inclusive
* Has a body mass index (BMI) between 18 and 32 kg/m2, inclusive
* Is able and willing to abstain from nicotine, alcohol, methylxanthine-containing beverages or food (e.g., coffee, tea, colas, chocolate, energy drinks), poppy seeds, and grapefruit juice for 48 hours prior to admission and for the duration of the study
* Is in good health generally, as determined by medical history, physical examination, clinical laboratory evaluations, and 12-lead electrocardiogram (ECG) at Screening
* Is willing and able to perform all study procedures as physically possible
* If sexually active, is willing to use a condom during sexual intercourse with female partners and to have their female partners use an additional effective means of contraception (e.g., intrauterine device, coil, diaphragm plus spermicide, oral contraceptive) or to abstain from sexual intercourse if female partner is not surgically sterile by tubal occlusion (ligation or occluding device) or postmenopausal from time of initial admission to the research facility until their last study visit

Exclusion Criteria:

* Baseline systolic blood pressure < 100 mmHg
* Subjects with spontaneous orthostatic hypotension, including a systolic decline of > 20 or diastolic change of > 10 mmHg or heart rate increase of > 30 bpm
* Has renal insufficiency as determined by eGFR < 65 mL/min/1.73m2 using the revised Cockcroft-Gault calculation: (140 - age [y])
* body weight [kg] / 72 serum creatinine [mg/dL]
* Has anemia (Hb < 12.5 gm/dL)
* Has history of cardiac or vascular disease, including the following: Congenital heart disease; Hypertension or hypotension; Cerebrovascular disease; aortic insufficiency; Clinically significant atrial or ventricular arrhythmias; Cardiac valvular heart disease; Hypertrophic cardiomyopathy or other cardiomyopathy
* Has a Screening ECG showing any of the following: Resting heart rate < 45 or > 100 bpm; PR interval > 210 msec; P wave duration > 120 msec; QRS interval < 70 or > 120 msec; Corrected QTc > 440 msec; QRS axis outside the range of -30 + 100 degrees; Right or left atrial enlargement or ventricular hypertrophy; Second- or third-degree atrioventricular block
* Heart block or intraventricular conduction defect
* Has diabetes mellitus Type I or Type II
* Is being treated with angiotensin-converting enzyme inhibitors, antihypertensive medications, diuretics, calcium-channel blockers, beta-blockers, cardiac glycosides, systemic anticholinergic agents, or drugs that may impair or enhance compensatory tachycardia
* Is being treated with growth hormone, insulin-like growth factor 1 (IGF-1), or anabolic steroids.
* Has any acute illness associated with volume dehydration (e.g., nausea/vomiting/diarrhea).
* Uses of any prescription medications, over-the-counter medications, or nutritional supplements within 10 days prior to dosing.
* Uses any other investigational product or investigational medical device within 90 days prior to screening or requires any investigational agent prior to completion of all scheduled study assessments.
* Consumes at least 14 units/week of alcohol (1 unit approximates 360 mL beer, 100 mL wine, or 35 mL spirits) or has significant history of alcoholism or drug/chemical abuse as determined by the Investigator.
* Has donated > 50 mL of blood or plasma within 60 days prior to study treatment administration.
* Has a positive urine drug screen or alcohol breath test result during Screening or upon admission to the research facility.
* Has used nicotine or tobacco-containing products (snuff, chewing tobacco, cigarettes,cigars, pipes, and nicotine replacements) within 90 days of the first dose of study treatment as confirmed by urine cotinine screen.
* Has a positive cotinine test result during Screening or upon admission to the research facility.
* Has a history of any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, hematological, or other major disorders as determined by the Investigator.
* Has had a clinically significant illness within 4 weeks of administration of the first dose of study treatment as determined by the Investigator.
* Is being treated with a concomitant medication that prolongs the QT/QTc interval within 7 days or 3 half-lives, whichever is longer, prior to the Screening Visit.
* Has AST or ALT greater than 3xULN or total bilirubin greater than 2xULN.
* Has known hypersensitivity to BMN 111 or its excipients.
* Has partner planning to become pregnant at any time during the study.
* Has any condition that, in the view of the Investigator, places the subject at high risk of poor treatment compliance or of not completing the study.

Ages: 22 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety based on vitals signs | Daily throughout the study Assessed for approximately 8 days following each single dose in Part 1, and for approximately 24 days following each daily dose in Part 2
Safety based on adverse events | Daily throughout the study Assessed for approximately 8 days following each single dose in Part 1, and for approximately 24 days following each daily dose in Part 2

SECONDARY OUTCOMES:
Pharmacokinetics | Daily on dosing days Assessed during Part 1 for approximately 10 days and during Part 2 for approximately 24 days
Safety based on cardiovascular effects | Daily throughout the study Assessed for approximately 8 days following each single dose in Part 1, and for approximately 24 days following each daily dose in Part 2

CONTACTS AND LOCATIONS:
Locations (1):
- Covance CRU Inc., Evansville, Indiana, United States